CLINICAL TRIAL: NCT06294262
Title: A Single-center, Observer-blind Study to Evaluate Safety, Immunogenicity, and Immunological Mechanisms of TETRALITE Influenza Vaccine With LiteVax Adjuvant, in Healthy Participants Aged 60 Years and Older and 18 to 50 Years.
Brief Title: Safety, Tolerability, Immunogenicity and Immunological Mechanisms of TETRALITE, a Novel Seasonal Influenza Vaccine
Acronym: TETRALITE-Ib
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LiteVax BV (Industry)
Collaborators: University Hospital, Ghent (Other); HarmonyCR, Melle, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023-508230-33-00
Record Dates: First submitted 2024-01-24; First posted 2024-03-05 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-05

CONDITIONS: Vaccination Reaction
Keywords: Vaccine adjuvant; LiteVax Adjuvant; Influenza virus vaccine; Seasonal influenza virus
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- VaxigripTetra in healthy adults aged 18-50 years (Active Comparator): A single, 0.5 mL intramuscular injection of VaxigripTetra without adjuvant in healthy adults aged 18-50 years (N = 12)
  Interventions: Biological: TETRALITE
- VaxigripTetra with 0.5 mg of LiteVax Adjuvant in healthy adults aged 18-50 years (Experimental): A single, 0.55 mL intramuscular injection of VaxigripTetra with 0.5 mg of LiteVax Adjuvant in healthy adults aged 18-50 years (N = 12)
  Interventions: Biological: TETRALITE
- VaxigripTetra with 1 mg of LiteVax Adjuvant in healthy adults aged 18-50 years (Experimental): A single, 0.55 mL intramuscular injection of VaxigripTetra with 1 mg of LiteVax Adjuvant in healthy adults aged 18-50 years (N = 12)
  Interventions: Biological: TETRALITE
- VaxigripTetra in healthy adults aged 60 years or older (Active Comparator): A single, 0.5 mL intramuscular injection of VaxigripTetra without adjuvant in healthy adults aged 60 years or older (N = 16)
  Interventions: Biological: TETRALITE
- VaxigripTetra with 0.5 mg of LiteVax Adjuvant in healthy adults aged 60 years or older (Experimental): A single, 0.55 mL intramuscular injection of VaxigripTetra with 0.5 mg of LiteVax Adjuvant in healthy adults aged 60 years or older (N = 16)
  Interventions: Biological: TETRALITE
- VaxigripTetra with 1 mg of LiteVax Adjuvant in healthy adults aged 60 years or older (Experimental): A single, 0.55 mL intramuscular injection of VaxigripTetra with 1 mg of LiteVax Adjuvant in healthy adults aged 60 years or older (N = 16)
  Interventions: Biological: TETRALITE

INTERVENTIONS:
Biological: TETRALITE — Intramuscular injection of VaxigripTetra with or without LiteVax Adjuvant
  Other Names: VaxigripTetra; LiteVax Adjuvant

SUMMARY:
The effect of LiteVax Adjuvant supplemented to licensed seasonal influenza vaccine on safety and immunogenicity will be investigated in both younger and older healthy participants. Local and systemic adverse events, and humoral and cellular immune responses will be determined at different time intervals after a single administration. Mode of action of LiteVax Adjuvant will examined by detailed genetic analysis and omics approaches such as transcriptomics, proteomics and metabolomics.

DETAILED DESCRIPTION:
The primary objective of this Phase 1b study is to evaluate the safety and tolerability of TETRALITE in participants aged 60 years and older and in participants aged 18 to 50 years. For this purpose, local and solicited Adverse Events (AEs), unsolicited AEs, and serious AEs, potential immune-mediated disease (pIMDs) and AEs of special interest (AESIs) will be assessed. For 7 days after vaccination, solicited local and systemic AEs will be recorded in a diary. Unsolicited AEs will be monitored for 28 days after vaccination. SAEs, pIMDs and AESIs will be assessed for 180 days after vaccination.

The secondary endpoints pertain to immunogenicity and include HI and MN titres. The HI antibody titers and MN antibody titers against the 4 vaccine influenza strains 7, 28 and 180 days after vaccination will be examined and compared to pre-vaccine levels. The current study aims to assess whether a dose level of 0.5 mg LVA and 1 mg LVA added to a standard dose of 15 µg of VaxigripTetra is capable of inducing a strong immune response, which could potentially translate into a higher vaccine effectiveness, especially in adults aged 60 years and older compared to adults aged 18 to 50 years. The increased susceptibility to influenza and other infectious diseases in adults aged 60 years and older is in part related to immunosenescence. Over time, the effectiveness of the immune system decreases. In general, vaccines are less immunogenic and reactogenic in the elderly compared to children or adults aged 18 to 50 years. Strategies to improve the immunogenicity in older adults include increasing the dose of antigen or adding an adjuvant.

The exploratory objectives include an evaluation of the mechanism(s) of (dose-dependent) action of LiteVax Adjuvant by using a systems vaccinology approaches including techniques to define genomic, transcriptomic, proteomic, metabolomic and lipidomic profiles and their interactions.

For this, blood samples will be collected in PAXgene tubes at Day 1 (pre-vaccination) 2 and 8. The analyses include differential gene expression and pathway analysis. The early timepoints will provide information on genes that are expressed at any given timepoint after vaccination compared to baseline. Additionally, genes that are differentially expressed in the adjuvanted vaccine group compared to the non-adjuvanted vaccine group will provide information on LiteVax Adjuvant. Finally, pathway enrichment will be performed. Given a list of differentially expressed genes, it will be determined how these genes work together, and which biological pathways are activated to induce antibody production.

ELIGIBILITY:
Inclusion Criteria:

1. Written signed informed consent obtained before any study-related activities.
2. Aged 18 to 50 years inclusive, at the time of signing the ICF in the younger age cohorts (Cohort 1, Cohort 2 and Cohort 3) and aged 60 years or older, at the time of signing the ICF in the older age cohorts (Cohort 4, Cohort 5 and Cohort 6).
3. Participants who are considered to be in good general health as determined by medical evaluation including medical history, physical examination (PE) and laboratory tests within 21 days prior to enrollment.
4. Participants with a BMI within the range 18.5 to 35 kg/m2 inclusive at screening.
5. Women who are not pregnant or breastfeeding, and one of the following conditions applies

   * Women of non-childbearing potential (WONCBP) as defined in Appendix 1. or
   * WOCBP and using a highly effective contraceptive method (with a failure rate of less than 1 % per year) as defined and described in Appendix 1 from at least 1 month prior to study vaccination and for 3 months post-vaccination. The investigator should evaluate the potential for contraceptive method failure (e.g. noncompliance, recently initiated) in relationship to study vaccination. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant. The participant should commit her abstinence to at least 1 month prior to study vaccination and for 3 months post-vaccination. If the participant will not maintain abstinence and changes her status, the participant must first commit to another highly effective method of contraception, which should be discussed with the investigator prior to terminating sexual abstinence as contraceptive method (34).
6. WOCBP must have a negative serum pregnancy test at screening and a negative urine pregnancy test before vaccination at Day 1. Refer to Section 8.3.5 for Pregnancy Testing. The investigator is responsible for review of medical history and menstrual history to decrease the risk for inclusion of a woman with an early undetected pregnancy.
7. Participants who are willing and able to comply with the study procedures and are in the view of the investigator capable of completing the study.

Exclusion Criteria:

Medical Conditions

1. History of previous laboratory confirmed influenza infection in the past 6 months, excluding laboratory confirmed COVID-19 infections, prior to the day of study vaccination.
2. Positive (in the past, suspected or ongoing) for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, and human immunodeficiency virus (HIV) antibody.
3. Past or current history of immune-mediated and/or autoimmune diseases as indicated by the investigator, e.g. diabetes mellitus type I and thyroid disease.
4. Serious reactions to vaccines that preclude receipt of study vaccinations as determined by the investigator.
5. Clinical conditions representing a contraindication for IM administration, as judged by the investigator, e.g. history of bleeding disorder (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM administration or blood draws.
6. History of confirmed hypersensitivity, allergy and/or anaphylaxis to eggs (ovalbumin or chicken proteins), squalene-based adjuvants, or other components of the study vaccine (neomycin, formaldehyde or octoxinol-9).
7. Current history of uncontrolled medical illness (unstable for the past 3 months) as judged by investigator, e.g. hypertension, diabetes mellitus type 2.
8. Past or current history of any neurological disorder, e.g. Guillain-Barré syndrome and seizure disorder other than: 1) childhood febrile seizures, or 2) seizures that have not required treatment within the last 3 years.
9. History of asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
10. Active malignancy or malignancy within the past 5 years, except basocellular carcinoma (single lesion) that has been fully removed.
11. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past 2 years or that is expected to require the use of oral or intravenous corticosteroids.
12. History of hereditary angioedema, acquired angioedema or idiopathic forms of angioedema.
13. History of idiopathic urticaria within the past year.
14. Current or recent (< 2 years ago) heavy smoking (> 20 cigarettes per day). If candidate stopped smoking > 2 years ago, the investigator will make an individual judgement based on the total packs per year and the candidate's overall health status. Drug - or alcohol abuse/addiction (including alcohol dependence), or psychiatric condition (e.g. past or present psychoses; disorder requiring lithium; or within 5 years prior to administration of study vaccine, a history of suicide plan or attempt), which in the investigator's opinion could compromise the participant's safety and/or compliance with the protocol.
15. A rash, dermatological condition or tattoos that would, in the opinion of the investigator, interfere with injection local reaction rating.

    Prior/Concomitant Therapy
16. Prior receipt of an investigational or licensed seasonal or pandemic influenza vaccine in the 9 months before administration of study vaccine or planning to receive the influenza vaccination during the study period.
17. Prior receipt of a live attenuated vaccine in the 28 days prior to administration of study vaccine, or within 14 days for subunit or inactivated vaccines other than seasonal or pandemic influenza vaccination, excluding COVID-19 vaccine.
18. Prior receipt of vaccination with TETRALITE + 0.5 mg LVA or TETRALITE + 2 mg LVA.
19. Prior receipt of COVID-19 vaccine in the 7 days before administration of study vaccine, or planning to receive a COVID-19 vaccine during the first 14 days following study vaccination.
20. Planning to receive a vaccine during the first 28 days following the administration of study vaccine, other than COVID-19 vaccine.
21. Currently participating in another clinical study, or planning to participate in another study during the study period, or administration of any investigational drug, vaccine or medical device in the 4 weeks prior to study vaccination (with the exception of influenza vaccine, refer to exclusion criterium 16).
22. Prior receipt of blood, blood-derived products or immunoglobulins in the 6 months prior to administration of study vaccine, or planning to receipt such product during the study period.
23. Chronic administration (defined as 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to vaccination or planned administration during the study (excluding topical, inhaled and intranasal preparations and intra-articular injections). For corticosteroids, this is prednisone >= 20 mg/day, or equivalent.
24. Current intake of more than 1 anticoagulant medication (coumarin derivatives, low molecular weight heparin, DOAC) or 1 anticoagulant medication in combination with antiaggregation medication.
25. Current anti-tuberculosis prophylaxis or therapy.
26. Elective surgery planned in the first 14 days following study vaccination. Other Exclusion Criteria
27. WOCBP who are pregnant, breast-feeding or planning to become pregnant during the study.
28. Participants with history of any medical conditions that, in opinion of the investigator, might interfere with the results of the study or pose additional risk to the participants due to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Characterise local and systemic AEs, and SAEs, pIMDs and AESIs to TETRALITE | 180 days
  Occurrence of solicited local and systemic AEs for 7 days, unsolicited AEs for 28 days, and SAEs, potential immune-mediated diseases (pIMDs), and adverse events of special interest (AESIs) for 180 days after vaccination. Local AEs include pain, redness, induration and swelling at the injection site. Systemic AEs include fever, headache, fatigue, myalgia, arthralgia, and malaise.
Characterise clinical hematology and biochemistry to TETRALITE | 28 days
  Occurrence of clinically abnormal hematology and serum biochemistry laboratory values 1 day, 7 days, and 28 days after vaccination versus baseline (Day 1, pre-vaccination). Hematology parameters include platelet count, red blood cell count (corpuscular volume, corpuscular haemoglobin and % reticulocytes), white blood cell counts (neutrophils, lymphocytes, monocytes, eosinophils, and basophils), haemoglobin and hematocrits. Biochemistry parameters include urea, creatinine, C-reactive protein, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, bilirubin, and high sensitive C-reactive protein.

SECONDARY OUTCOMES:
Characterise HI antibody response to the four vaccine strains of TETRALITE in serum | 180 days
  The HI antibody titers against the 4 vaccine influenza strains in serum samples 7 days, 28 days, and 180 days after vaccination versus baseline (Day 1, pre-vaccination).
Characterise MN antibody response to the four vaccine strains of TETRALITE in serum | 180 days
  The microneutralization (MN) antibody titers against the 4 vaccine influenza strains in serum samples 7 days, 28 days, and 180 days after vaccination versus baseline (Day 1, pre-vaccination).

OTHER OUTCOMES:
Characterise mechanisms of action of LiteVax Adjuvant | 28 days
  Characterization of gene transcription induced by vaccination by examining differentially expressed genes, and enriched pathways at baseline (Day 1, pre-vaccination), Day 2, and Day 8, and changes occurring between Day 2 and baseline, Day 8 and baseline, and Day 8 and Day 2.
  Characterization of the innate immune response and its dynamics after vaccination by examining the differentially expressed genes and enriched pathways at baseline (Day 1, pre-vaccination), Day 2, and Day 8, and changes occurring between Day 2 and baseline, Day 8 and baseline, and Day 8 and Day 2.
  Characterization of (activated) cells, cell clusters or cell states and identification of expressed genes, and changes in gene expression levels in each cell type at baseline (Day 1, pre-vaccination), Day 2, and Day 8, and changes occurring between Day 2 and baseline, Day 8 and baseline, and Day 8 and Day 2.
Characterise T-cell responses to TETRALITE in PBMCs | 180 days
  T cell mediated immune response in peripheral blood mononuclear cells (PBMCs) 7 days and 180 days after vaccination versus baseline (Day 1, pre-vaccination) as confirmed by the presence of influenza-specific CD4+ and CD8+ T cells producing at least CD40L, IL-2, IFNγ and/or TNFα as measured by flow cytometry (intracellular cytokine staining).
Characterise B-cell response to TETRALITE in PBMCs | 180 days
  B cell response in PBMCs 7 days and 180 days after vaccination versus baseline (Day 1, pre-vaccination), as confirmed by the presence of plasmablasts as measured by ELISPOT
Characterise molecular features of vaccine-induced immunity by RNA sequencing | 180 days
  Assays may include but are not limited to RNA sequencing of RNA extracted from whole blood (bulk) and from PBMCs (single cell).
Characterise antibody response to influenza virus antigens other than hemaglutunin of the vaccine strains of TETRALITE | 180 days
  Assays may include but are not limited to antibody responses against neuraminidase, nucleoprotein and matrix protein.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Gent, Ghent, Belgium